CLINICAL TRIAL: NCT02260882
Title: A Study Evaluating the Safety and Immunogenicity of Revaccination With 23-Valent Pneumococcal Polysaccharide Vaccine in Older Japanese Adults
Brief Title: Revaccination With PNEUMOVAX™ 23 in Older Japanese Adults (V110-902)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V110-902; 152859 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Pneumococcal Infection
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Revaccination Group (Experimental): 0.5 mL intramuscular injection (deltoid or lateral mid-thigh) of PNEUMOVAX™ 23 vaccine on Day 1 for participants who received an initial vaccination at least 5 years prior
  Interventions: Biological: PNEUMOVAX™ 23
- Primary Vaccination Group (Experimental): 0.5 mL intramuscular injection (deltoid or lateral mid-thigh) of PNEUMOVAX™ 23 vaccine on Day 1 for participants who have never received PNEUMOVAX™ 23 vaccination
  Interventions: Biological: PNEUMOVAX™ 23

INTERVENTIONS:
Biological: PNEUMOVAX™ 23 — PNEUMOVAX™ 23 (23-Valent Pneumococcal Polysaccharide Vaccination, V110, PPV23)

SUMMARY:
The purpose of this study is to determine if revaccination with pneumococcal vaccine (PNEUMOVAX™ 23, V110) is well tolerated and produces an immune response in older Japanese adults. The primary hypothesis being tested is that the geometric mean concentration of antibodies to pneumococcal polysaccharide serotypes 3, 6B, and 23F at 4 weeks after revaccination will be superior to that before revaccination in Japanese adults who received a primary vaccination at least 5 years before revaccination.

ELIGIBILITY:
Inclusion Criteria:

* Japanese participant
* Good health or any underlying chronic illness is documented to be in stable condition
* Revaccination Group: received one documented PNEUMOVAX™ 23 vaccination at least 5 years before enrollment in the study
* Primary Vaccination Group: no prior history with PNEUMOVAX™ 23 vaccination Exclusion Criteria:
* Known allergy or sensitivity to any of the components of the study vaccine
* History of pneumococcal conjugate vaccination
* Known or suspected immune dysfunction, immunosuppression, or autoimmune disease. Participants with a history of cancer who are not actively treated and not immunosuppressed will be eligible
* Functional or anatomic asplenia
* Received immunoglobulin within 6 months before study vaccine or is planned during the study
* Received any investigational drugs or vaccines within 2 months before study vaccination
* History of pneumococcal disease (positive culture from blood or other normally sterile site)
* Thrombocytopenia or any coagulation disorder that would contraindicate intramuscular injection
* History of convulsion
* Previously diagnosed with immunodeficiency or has a close relative with congenital immune deficiency
* Participating in any other clinical trial

Ages: 70 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 243 (Actual)
Dates: Start 2014-10-31 (Actual); Primary Completion 2015-04-09 (Actual); Study Completion 2015-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Kawakami K, Kishino H, Kanazu S, Toshimizu N, Takahashi K, Sterling T, Wang M, Musey L. Revaccination with 23-valent pneumococcal polysaccharide vaccine in the Japanese elderly is well tolerated and elicits immune responses. Vaccine. 2016 Jul 19;34(33):3875-81. doi: 10.1016/j.vaccine.2016.05.052. Epub 2016 Jun 10. PMID 27265450

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Depending on prior history of Pneumovax™ 23 vaccination, 161 participants with a history of prior Pneumovax™ 23 vaccination were enrolled into the Revaccination group and 82 participants without a history of prior Pneumovax™ vaccination were enrolled into the Primary vaccination group.
Period: Overall Study
Arm/Group | Revaccination Group | Primary Vaccination Group
Started | 161 | 82
Completed | 161 | 81
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: One participant in the Primary Vaccination Group was withdrawn from the study before vaccination because of a protocol violation. Baseline Characteristics are based on the Full Analysis Set: participants who received at least one vaccination.
Groups:
- Total: Total of all reporting groups
Arm/Group | Revaccination Group | Primary Vaccination Group | Total
Number analyzed (Participants) | 161 | 81 | 242
Age, Continuous [Mean (Standard Deviation); unit: Years] | 78.8 (4.8) | 78.2 (5.0) | 78.6 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 46 | 140
  Male | 67 | 35 | 102

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Serotype-Specific Antibody Geometric Mean Concentration at 4 Weeks After Revaccination
Description: Serum antibodies to pneumococcal serotypes were measured by enzyme-linked immunosorbent assays. Geometric mean antibody concentrations (GMCs) were calculated at Baseline and 4 weeks postvaccination. Geometric Mean Fold Rise was the GMC at 4 weeks after vaccination minus the GMC at Baseline.
Time Frame: Baseline and 4 weeks after revaccination
Population: Per Protocol Set: all participants in the Revaccination Group except those with a protocol deviation, including those with blood collection outside the protocol-specified window.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Fold Rise
Arm/Group | Revaccination Group
Number analyzed (Participants) | 161
Geometric Mean Fold Rise
  Serotype 3: n=161 | 2.72 [2.35 to 3.14]
  Serotype 6B: n=161 | 2.27 [2.02 to 2.55]
  Serotype 23F: n=160 | 2.40 [2.12 to 2.72]
Statistical Analysis 1: Comparison: Revaccination Group; Serotype 3. The statistical success criterion for demonstrating greater geometric mean antibody concentrations at 4 weeks postvaccination is that the lower bound of the 2-sided 95% confidence interval in Geometric Mean Fold Rise will be greater than 1 for all 3 serotypes; Test type: Superiority or Other; p < 0.001, t-test, 1 sided
Statistical Analysis 2: Comparison: Revaccination Group; Serotype 6B. The statistical success criterion for demonstrating greater geometric mean antibody concentrations at 4 weeks postvaccination is that the lower bound of the 2-sided 95% confidence interval in Geometric Mean Fold Rise will be greater than 1 for all 3 serotypes; Test type: Superiority or Other; p < 0.001, t-test, 1 sided
Statistical Analysis 3: Comparison: Revaccination Group; Serotype 23F. The statistical success criterion for demonstrating greater geometric mean antibody concentrations at 4 weeks postvaccination is that the lower bound of the 2-sided 95% confidence interval in Geometric Mean Fold Rise will be greater than 1 for all 3 serotypes; Test type: Superiority or Other; p < 0.001, t-test, 1 sided

2. Secondary Outcome: Change From Baseline in Serotype-Specific Antibody Geometric Mean Concentration at 4 Weeks After Primary Vaccination
Description: as for outcome 1
Time Frame: Baseline and 4 weeks after primary vaccination
Population: Per Protocol Set: all participants in the Primary Vaccination Group except those with a protocol deviation, including those with blood collection outside the protocol-specified window
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Fold Rise
Arm/Group | Primary Vaccination Group
Number analyzed (Participants) | 81
Geometric Mean Fold Rise
  Serotype 3 | 4.01 [3.17 to 5.08]
  Serotype 6B | 5.83 [4.41 to 7.69]
  Serotype 23F | 6.11 [4.65 to 8.02]

3. Secondary Outcome: Percentage of Participants With an Adverse Event of Injection-site Erythema
Description: An adverse event is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product. Percentage of participants with an adverse event of injection-site erythema recorded on the Vaccine Report Card (VRC) during the first 5 days after vaccination was recorded.
Time Frame: Up to 5 days after vaccination
Population: All Subjects as Treated set: all participants who received study vaccine.
Measure: Number; unit: Percentage of participants
Arm/Group | Revaccination Group | Primary Vaccination Group
Number analyzed (Participants) | 161 | 81
Percentage of participants | 35.4 | 14.8

4. Secondary Outcome: Percentage of Participants With an Adverse Event of Injection-site Swelling
Description: An adverse event is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product. Percentage of participants with an adverse event of injection-site swelling recorded on the VRC during the first 5 days after vaccination was recorded.
Time Frame: Up to 5 days after vaccination
Population: All Subjects as Treated set: all participants who received study vaccine.
Measure: Number; unit: Percentage of participants
Arm/Group | Revaccination Group | Primary Vaccination Group
Number analyzed (Participants) | 161 | 81
Percentage of participants | 38.5 | 17.3

5. Secondary Outcome: Percentage of Participants With an Adverse Event of Injection-site Pain
Description: An adverse event is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product. Percentage of participants with an adverse event of injection-site pain recorded on the VRC during the first 5 days after vaccination was recorded.
Time Frame: Up to 5 days after vaccination
Population: All Subjects as Treated set: all participants who received study vaccine.
Measure: Number; unit: Percentage of participants
Arm/Group | Revaccination Group | Primary Vaccination Group
Number analyzed (Participants) | 161 | 81
Percentage of participants | 62.7 | 46.9

6. Secondary Outcome: Percentage of Participants With an Adverse Event of Pyrexia
Description: Percentage of participants with an adverse event of pyrexia (>=37.5°C, oral) recorded on the VRC during the first 5 days after vaccination was recorded.
Time Frame: Up to 5 days after vaccination
Population: All Subjects as Treated set: all participants who received study vaccine.
Measure: Number; unit: Percentage of participants
Arm/Group | Revaccination Group | Primary Vaccination Group
Number analyzed (Participants) | 161 | 81
Percentage of participants | 6.8 | 1.2

7. Secondary Outcome: Percentage of Participants With an Adverse Event of Myalgia
Description: An adverse event is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product. Percentage of participants with an adverse event of myalgia recorded on the VRC during the first 14 days after vaccination was recorded.
Time Frame: Up to 14 days after vaccination
Population: All Subjects as Treated set: all participants who received study vaccine.
Measure: Number; unit: Percentage of participants
Arm/Group | Revaccination Group | Primary Vaccination Group
Number analyzed (Participants) | 161 | 81
Percentage of participants | 0.0 | 0.0

8. Secondary Outcome: Percentage of Participants With an Adverse Event of Arthralgia
Description: An adverse event is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product. Percentage of participants with an adverse event of arthralgia recorded on the VRC during the first 14 days after vaccination was recorded.
Time Frame: Up to 14 days after vaccination
Population: All Subjects as Treated set: all participants who received study vaccine.
Measure: Number; unit: Percentage of participants
Arm/Group | Revaccination Group | Primary Vaccination Group
Number analyzed (Participants) | 161 | 81
Percentage of participants | 0.0 | 0.0

9. Secondary Outcome: Percentage of Participants With an Adverse Event of Headache
Description: An adverse event is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product. Percentage of participants with an adverse event of headache recorded on the VRC during the first 14 days after vaccination was recorded.
Time Frame: Up to 14 days after vaccination
Population: All Subjects as Treated set: all participants who received study vaccine.
Measure: Number; unit: Percentage of participants
Arm/Group | Revaccination Group | Primary Vaccination Group
Number analyzed (Participants) | 161 | 81
Percentage of participants | 1.9 | 1.2

10. Secondary Outcome: Percentage of Participants With an Adverse Event of Fatigue
Description: An adverse event is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product. Percentage of participants with an adverse event of fatigue recorded on the VRC during the first 14 days after vaccination was recorded.
Time Frame: Up to 14 days after vaccination
Population: All Subjects as Treated set: all participants who received study vaccine.
Measure: Number; unit: Percentage of participants
Arm/Group | Revaccination Group | Primary Vaccination Group
Number analyzed (Participants) | 161 | 81
Percentage of participants | 1.2 | 0.0

ADVERSE EVENTS:
Time Frame: All adverse events: up to 14 days after vaccination; deaths and vaccine-related serious adverse events: up to 36 days after vaccination
Arm/Group | Revaccination Group | Primary Vaccination Group
Serious Adverse Events (participants affected / at risk) | 4/161 | 0/81
Other Adverse Events (participants affected / at risk) | 113/161 | 41/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Revaccination Group (N=161) | Primary Vaccination Group (N=81)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Herpes virus infection (Infections and infestations) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Revaccination Group (N=161) | Primary Vaccination Group (N=81)
Injection-site erythema (General disorders) | 57 (57) | 12 (12)
Injection-site pain (General disorders) | 101 (102) | 38 (38)
Injection-site pruritus (General disorders) | 11 (11) | 2 (2)
Injection-site swelling (General disorders) | 62 (62) | 14 (14)
Pyrexia (General disorders) | 11 (11) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the trial without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial.